CLINICAL TRIAL: NCT06214923
Title: Neural Mechanisms of Immersive Virtual Reality in Chronic Pain
Brief Title: Neural Mechanisms of Immersive Virtual Reality in Chronic Pain (VR TMD EEG)
Acronym: VR TMD EEG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Luana Colloca, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HP-00095888 (VR TMD EEG)
Record Dates: First submitted 2023-12-18; First posted 2024-01-22 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Pain; Virtual Reality; Placebo; Temporomandibular Disorder
Keywords: TMD volunteers; VR; Clinical Pain; Ecological Momentary Assessment
MeSH Terms: conditions — Pain; Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: This is a 2 (high- vs. low-impact pain) by 3 (3-week Active VR vs. 3-week Sham VR vs. 3-week NH) conditions mixed experimental design. TMD participants will be clinically phenotype into high-impact or low-impact pain groups according to Graded Chronic Pain Scale (GCPS). All participants will go through Active VR, Sham VR and NH phases (3-week each).
  There will be 4 in-person visits where participants will be monitored for changes in cortical excitability via PAF oscillations and clinical benefit via Ecological Momentary Assessments (EMA) during the 3-week conditions.
  Crossover Study Model was chosen because each participant will receive VR, Sham-VR, and No-VR in random order
Who Masked: Participant
Masking Description: Participants will be blinded to the VR and Sham-VR conditions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- High impact TMD (Other): Other: TMD Phenotype
  TMD participants will be clinically phenotyped into two between-subject groups based on their score on the Graded Chronic Pain Scale (GCPS). This group will have a GCPS grade 2b, 3, and 4.
  Interventions: Device: RelieVRx; Device: Sham-VR; Other: No-VR (natural history control)
- Low impact TMD (Other): Other: TMD Phenotype
  TMD participants will be clinically phenotyped into two between-subject groups based on their score on the Graded Chronic Pain Scale (GCPS). This group will have a GCPS grade 0, 1, and 2a
  Interventions: Device: RelieVRx; Device: Sham-VR; Other: No-VR (natural history control)

INTERVENTIONS:
Device: RelieVRx — Participants will use RelieVRx daily for 20min/day for 3 weeks
  Other Names: Active-VR
Device: Sham-VR — Participants will use Sham-VR, consisting of video, images, and sound in a head-mounted display but lack the "sense of presence" and immersive features of Active-VR (for example, scene changes with head movement). Participants will use the Sham-VR daily for 20min/day for 3 weeks
Other: No-VR (natural history control) — Participants will continue regular/usual care without any VR devices (goggles or audiovisual input)

SUMMARY:
This project examines, in chronic pain, the mechanisms of immersive virtual reality compared to the mechanisms of placebo hypoalgesia. The potential of developing new non-pharmacological premises for low-risk interventions for pain management is high.

DETAILED DESCRIPTION:
Virtual reality (VR) has been seen as an intervention for alleviating clinical chronic (and acute) pain. An approach to pain management utilizing VR presents opportunities for reducing pain and suffering by using immersive, aesthetic, and multisensory stimulation. Investigator will analyze the behavioral and neural mechanisms of active VR against sham VR as two methods that investigate descending pain modulation. Thus, the central hypothesis is that those who respond to placebos will likely respond to active VR. If VR-induced analgesia depends upon the release of endogenous opioids.

In this project, the investigators will determine the effects of VR at the neural and clinical levels directly for TMD participants, inviting participants from an existing Colloca Lab-based cohort phenotyped for diagnosis, grade, and low/high impact pain profiles and prospective TMD participants in collaboration with Johns Hopkins University. These participants have agreed to be recontacted for further research.

In this study, based on our PAF study and modulation of autonomic measurements via VR, we will determine the role of acute and 3-week VR intervention to help restore PAF oscillations to normal. PAF and autonomic measurements will be collected in TMD participants characterized by low/high-impact pain. All participants will go through Active VR, Sham VR and NH phases (3-week each) where participants will be monitored for changes in cortical excitability via PAF oscillations and clinical benefit via EMA.

ELIGIBILITY:
Inclusion Criteria:

* Age (18-88 years)
* English speaker (written and spoken)
* Temporal Mandibular Disorder (TMD) for at least 3 months
* TMD Grade Chronic Pain Scale (GCPS) ≥ 0

Exclusion Criteria:

* Present or past degenerative neuromuscular disease
* Cardiovascular, neurological diseases, pulmonary abnormalities, kidney disease, liver disease, history of cancer within past 3 years
* Cervical pain (e.g. stenosis, radiculopathy)
* Any personal (or family first degree) history of mania, schizophrenia, or other psychoses
* Severe psychiatric condition (e.g. schizophrenia, bipolar disorders, autism) leading to hospitalization within the last 3 years.
* Use of Antipsychotics (e.g., Risperdal, Ability and clozaril)Lifetime alcohol/drug dependence or alcohol/drug abuse in past 3 months
* Pregnancy or breast feeding
* Color-blindness
* Impaired or uncorrected hearing
* Non-dominant hand
* Any facial trauma that has occurred in the last 6 weeks
* History of a severe facial trauma in the last 2-3 months
* Conditions that would interfere with the VR mask placement (e.g. trauma, burn, infection)
* Known history of severe motion sickness
* Non-removable head cover, artificial hair, certain types of braids or dreadlocks
* History of fainting
* History of angioedema
* Failed drug test (testing for opiates, cocaine, methamphetamines, and amphetamines)

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Peak alpha frequency (PAF) | We will acquire 2-10 min of baseline EEG with open eyes and 2-10 min of EEG with closed eyes. This measurement will occur at each of the four in-person visit approximately every 3 weeks.
  EEG response PAF when participants are undergoing the in-person VR
Objective incremental Celsius changes in heat-pain tolerance | The heat incremental changes range from 30 sec to 2 min tolerance. This measurement will occur at each of the four in-person visit approximately every 3 weeks.
  Heat pain tolerance to incremental change in temperature will be obtained using a timer (minutes of tolerance)

SECONDARY OUTCOMES:
Subjective VAS (Visual Analog Scale) scores for mood, situational anxiety, and pain intensity/unpleasantness | Daily during the 3-week condition timeframe
  Participants will take Ecological Momentary Assessment questionnaires. Minimum Value: 0 Maximum Value: 100 Score interpretation: 0=not at all, 100=most/strongest For example, anxiety on a scale of 0-100, 0=no anxiety, 100=the most anxious

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Luana Colloca, Baltimore, Maryland
  - University of Maryland, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No
At this time, there is neither intent nor plan to share IPD.

REFERENCES:
- [Background] Honzel E, Murthi S, Brawn-Cinani B, Colloca G, Kier C, Varshney A, Colloca L. Virtual reality, music, and pain: developing the premise for an interdisciplinary approach to pain management. Pain. 2019 Sep;160(9):1909-1919. doi: 10.1097/j.pain.0000000000001539. No abstract available. PMID 30817437
- [Background] Colloca L, Raghuraman N, Wang Y, Akintola T, Brawn-Cinani B, Colloca G, Kier C, Varshney A, Murthi S. Virtual reality: physiological and behavioral mechanisms to increase individual pain tolerance limits. Pain. 2020 Sep 1;161(9):2010-2021. doi: 10.1097/j.pain.0000000000001900. PMID 32345915
- [Background] Amanzio M, Benedetti F. Neuropharmacological dissection of placebo analgesia: expectation-activated opioid systems versus conditioning-activated specific subsystems. J Neurosci. 1999 Jan 1;19(1):484-94. doi: 10.1523/JNEUROSCI.19-01-00484.1999. PMID 9870976
- [Background] Colloca L. The Placebo Effect in Pain Therapies. Annu Rev Pharmacol Toxicol. 2019 Jan 6;59:191-211. doi: 10.1146/annurev-pharmtox-010818-021542. Epub 2018 Sep 14. PMID 30216744